CLINICAL TRIAL: NCT06978218
Title: Cognitive Changes in Menopause: A Comparative Analysis of Brain Fog and Quality of Life
Brief Title: Brain Fog and Life Quality in Menopause
Status: Completed | Type: Observational
Sponsor: Merve Coskun (Other)
Responsible Party: Sponsor-Investigator, Merve Coskun, Assistant professor, Acibadem University
Organization: Acibadem University (Other)
Other Study IDs: 2025-06-251
Record Dates: First submitted 2025-05-08; First posted 2025-05-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Menopause; Cognitive Dysfunction; Memory Disorders; Quality of Life; Women's Health; Perimenopausal Disorder; Postmenopausal Symptoms
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This clinical study aims to investigate cognitive changes in women undergoing the menopausal transition, with a specific focus on the prevalence, characteristics, and impact of brain fog. The research will assess how declining estrogen levels influence cognitive domains such as memory, attention, and executive function across different menopausal stages (perimenopause, menopause, and postmenopause). Through a comparative and observational design, the study will evaluate the relationship between subjective cognitive complaints and menopause-specific quality of life. Findings are expected to inform the development of non-pharmacological strategies-such as lifestyle modifications and cognitive health interventions-to mitigate cognitive decline and improve overall well-being in midlife women.

DETAILED DESCRIPTION:
Menopause is a natural biological process characterized by a decline in ovarian function and a marked reduction in estrogen and progesterone levels, often accompanied by elevated follicle-stimulating hormone (FSH) levels. These hormonal changes are known to influence various physiological and psychological domains, including cognitive functioning. Recent evidence suggests that many women report subjective cognitive difficulties during the menopausal transition, commonly described as "brain fog," which includes symptoms such as forgetfulness, difficulty concentrating, slowed thinking, and word-finding problems.

This study is designed to systematically examine the nature and extent of cognitive changes during the menopausal transition, with a focus on comparing different stages-perimenopause, menopause, and postmenopause. Using validated cognitive screening tools and self-report measures, the study will assess domains including attention, memory, and executive function, and evaluate how these relate to menopause-specific quality of life.

In addition to cognitive assessments, participants will complete surveys addressing mood, sleep quality, physical activity, and perceived stress, as these are potential moderators or mediators of cognitive function during menopause. The study also aims to explore correlations between the severity of brain fog symptoms and demographic or lifestyle-related factors such as age, BMI, education level, and health behaviors.

By adopting a cross-sectional comparative approach, this research seeks to better characterize brain fog as a clinical concern in menopausal women and to identify vulnerable subgroups who may benefit from targeted cognitive and lifestyle interventions. The findings are expected to contribute to the growing body of knowledge on neuroendocrinology and women's brain health, and may support the development of tailored clinical guidelines or integrative care models for managing cognitive complaints during menopause.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 and 60 years.
* In any stage of menopause.
* Able to complete the Brain Fog Scale and Menopause-Specific Quality of Life Scale due to cognitive and physical capability.
* Willing to participate in the study voluntarily.
* Able to read and write in Turkish.

Exclusion Criteria:

* Diagnosed with neurological or psychiatric disorders (e.g., Alzheimer's, Dementia, Schizophrenia, etc.).
* Currently receiving hormone therapy.
* Experiencing menstrual irregularities due to reasons other than menopause.
* Unable to complete the scales due to visual impairment or significant cognitive limitations.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study is designed to evaluate the cognitive changes, brain fog, and quality of life specifically in women undergoing menopause. Therefore, only female participants who are currently experiencing or have experienced menopause are eligible to participate.
Study Population: The study population consists of women aged between 40 and 60 years who are experiencing or have experienced menopause. The participants will be selected from women at different stages of menopause, including peri-menopause, menopause, and post-menopause. The study aims to include a diverse group of women to understand the variations in cognitive changes and quality of life during different stages of menopause.
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Cognitive Function Changes and Severity of Brain Fog Symptoms (BFS) | At baseline (one-time assessment at enrollment)
  The primary outcome measure of this study is to assess changes in cognitive function and the severity of brain fog symptoms in women at different stages of menopause (peri-menopause, menopause, and post-menopause). The Brain Fog Scale allows participants to subjectively assess their brain fog symptoms, including forgetfulness, difficulty focusing, mental slowing, and trouble finding words. Measurement Content:
  Mental Fatigue: Feelings of mental tiredness and its impact on daily life.
  Impaired Cognitive Sharpness: Issues related to attention, memory, and cognitive clarity.
  Mental Cloudiness: Loss of mental clarity and difficulty organizing thoughts.
  Scoring System: The BFS uses a 5-point Likert scale (0: Never, 4: Always) to assess symptoms. Higher scores indicate more pronounced brain fog symptoms.
Menopause-Specific Quality of Life (MENQOL) | At baseline (one-time assessment at enrollment)
  The primary outcome measure of this study is to evaluate the impact of menopause on the overall quality of life (QOL) in women at different stages of menopause (peri-menopause, menopause, and post-menopause). The MENQOL assesses various aspects of life that are influenced by menopause, including physical, psychosocial, sexual, and vasomotor symptoms.The MENQOL uses a 7-point Likert scale, with scores ranging from 0 (no problem) to 6 (severe problem). Higher scores indicate greater severity of symptoms and a lower quality of life related to menopause.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Coşkun, Asst. Prof., Principal Investigator — Acibadem University
Locations (1):
- Merve Coşkun, Ataşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhu C, Thomas EH, Li Q, Arunogiri S, Thomas N, Gurvich C. Evaluation of the Everyday Memory Questionnaire-Revised in a menopausal population: understanding the brain fog during menopause. Menopause. 2023 Nov 1;30(11):1147-1156. doi: 10.1097/GME.0000000000002256. Epub 2023 Oct 2. PMID 37788429
- [Background] Shrividya, S., & Joy, M. (2021). Brain fog among perimenopausal women: A comparative study. Journal of International Women's Studies, 22(6), 11-21.
- [Background] Mosconi L, Rahman A, Diaz I, Wu X, Scheyer O, Hristov HW, Vallabhajosula S, Isaacson RS, de Leon MJ, Brinton RD. Increased Alzheimer's risk during the menopause transition: A 3-year longitudinal brain imaging study. PLoS One. 2018 Dec 12;13(12):e0207885. doi: 10.1371/journal.pone.0207885. eCollection 2018. PMID 30540774
- [Background] Bean, L. A., Ianov, L., & Foster, T. C. (2021). Estrogen receptors, the hippocampus, and memory: Neural systems approach to understanding estrogen function. Hormones and Behavior, 127, 104893.
- [Background] Bas M, Kahriman M, Gencalp C, Koseoglu SK, Hajhamidiasl L. Adaptation and Validation of the Turkish Version of the Brain Fog Scale. Int J Environ Res Public Health. 2024 Jun 14;21(6):774. doi: 10.3390/ijerph21060774. PMID 38929020
- [Background] Debowska, A., Boduszek, D., Ochman, M., Hrapkowicz, T., Gaweda, M., Pondel, A., & Horeczy, B. (2024). Brain Fog Scale (BFS): scale development and validation. Personality and Individual Differences, 216, 112427.
- [Background] Polit, D., & Beck, C. (2017). Nursing research : generating and assessing evidence for nursing practice (10th ed.). Lippincott Williams & Wilkins. ISBN 978-1-4963-0023-2, ss-380, 563-564
- [Background] Lee KS, Jung MS, Kim M, Cha K, Chung E. Impact of Cognitive Aging on Health-Related Quality of Life in Menopausal Women. Osong Public Health Res Perspect. 2020 Aug;11(4):185-193. doi: 10.24171/j.phrp.2020.11.4.07. PMID 32864309
- [Background] Gümüşay, M., & Erbil, N. (2019). Kadınların menopoza özgü yaşam kalitesine menopoz tutumunun etkisi. Ordu Üniversitesi Hemşirelik Çalışmaları Dergisi, 2(2), 96-109.
- [Background] Kuck MJ, Hogervorst E. Stress, depression, and anxiety: psychological complaints across menopausal stages. Front Psychiatry. 2024 Feb 22;15:1323743. doi: 10.3389/fpsyt.2024.1323743. eCollection 2024. PMID 38455517
- [Result] Maki PM, Jaff NG. Brain fog in menopause: a health-care professional's guide for decision-making and counseling on cognition. Climacteric. 2022 Dec;25(6):570-578. doi: 10.1080/13697137.2022.2122792. Epub 2022 Sep 30. PMID 36178170
- [Result] Maki PM, Jaff NG. Menopause and brain fog: how to counsel and treat midlife women. Menopause. 2024 Jul 1;31(7):647-649. doi: 10.1097/GME.0000000000002382. Epub 2024 Jun 17. PMID 38888619